CLINICAL TRIAL: NCT04420689
Title: Phase 1/2 Trial of ALM-488 in Patients Undergoing Head & Neck Surgery
Brief Title: Bevonescein to Highlight Nerves in Patients Undergoing Head & Neck Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alume Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ALM-488-001
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Parotid Neoplasm; Thyroid Neoplasms; Head and Neck Neoplasms; Surgery; Nerve Injury; Imaging
Keywords: Nerve; Fluorescence; Surgery; Imaging; Real-time; Intraoperative; Highlighting
MeSH Terms: conditions — Parotid Neoplasms; Thyroid Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/Phase 2 study in patients undergoing Head & Neck Surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation/De-Escalation Cohorts (Experimental): This arm of the study will include Dose Escalation/De-Escalation cohorts of Bevonescein (ALM-488).
  Interventions: Drug: Bevonescein
- Dose Timing Cohorts (Experimental): This arm of the study will include Dose Timing cohorts of Bevonescein (ALM-488).
  Interventions: Drug: Bevonescein

INTERVENTIONS:
Drug: Bevonescein — Bevonescein Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
  Other Names: ALM-488

SUMMARY:
Bevonescein to Highlight Nerves in Patients Undergoing Head & Neck Surgery

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and efficacy of Bevonescein (ALM-488) administered as an intravenous (IV) infusion to patients undergoing head & neck surgery. The study will also characterize the pharmacokinetics of Bevonescein (ALM-488) in this subject population and determine the dose of Bevonescein (ALM-488) needed to generate a fluorescence signal in nerve tissue to enable fluorescence recordings and image analysis with an imaging system. The study will also evaluate the effect of timing of Bevonescein (ALM-488) administration, relative to surgery, on fluorescence characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. A neoplasm located in the head and neck.
2. Primary surgical treatment is by parotidectomy, or thyroidectomy, or cervical neck dissection.
3. Can understand and is willing to sign a written informed consent document.
4. ≥18 years of age.
5. Life expectancy of at least 6 months.
6. Normal liver and kidney functions.
7. If of childbearing potential, must have a negative urine or serum pregnancy test and be using a medically acceptable form of contraception (e.g., hormonal birth control, intrauterine devices, double-barrier method) or abstinence. The subject, if male, must use a medically acceptable form of contraception (e.g. condom) or abstinence.
8. Plans to undergo head and neck surgery.

Exclusion Criteria:

1. Prior radiation or chemotherapy for any prior head and neck neoplasm.
2. Open surgery in the ipsilateral head and neck within 1 year.
3. Abnormal cardiac rhythm not controlled with medication, history of stroke, coronary events and/or heart failure within 1 year.
4. Current evidence of renal disease.
5. Pregnant or breastfeeding.
6. Unresolved acute toxicity from prior anti-cancer therapy.
7. History of fluorescein allergy.
8. Any other criteria deemed by the Principal Investigator that may prevent the patient from successfully completing the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Harvard-Mass Eye & Ear, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YJ, Orosco RK, Bouvet M, Richmon JD, Berman BJ, Crawford KL, Hom M, Nguyen QT, Rosenthal EL. Intraoperative nerve-specific fluorescence visualization in head and neck surgery: a Phase 1 trial. Nat Commun. 2025 Jul 2;16(1):6060. doi: 10.1038/s41467-025-60737-x. PMID 40595556

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Defining Cohort 100mg: This group of the study will receive 100mg of Bevonescein (ALM-488).
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue. 100mg of ALM-488 will be intravenously infused.
- Dose Defining Cohort 200mg: This group of the study will receive 200mg of ALM-488.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue. 200mg of ALM-488 will be intravenously infused.
- Dose Defining Cohort 400mg: This group of the study will receive 400mg of Bevonescein (ALM-488).
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue. 400mg of ALM-488 will be intravenously infused.
- Dose Defining Cohort 500mg: This group of the study will receive 500mg of Bevonescein (ALM-488).
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue. 500mg of ALM-488 will be intravenously infused.
- Dose Defining Cohort 600mg: This group of the study will receive 600mg of Bevonescein (ALM-488).
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue. 600mg of ALM-488 will be intravenously infused.
- Dose Timing Cohort 3-5 Hours: This arm of the study will include patients infused wtih Bevonescein (ALM-488) at 500mg 3-5 hours prior to skin incision.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing Cohort 1-3 Hours: This arm of the study will include patients infused wtih Bevonescein (ALM-488) at 500mg 1-3 hours prior to skin incision.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
Period: Overall Study
Arm/Group | Dose Defining Cohort 100mg | Dose Defining Cohort 200mg | Dose Defining Cohort 400mg | Dose Defining Cohort 500mg | Dose Defining Cohort 600mg | Dose Timing Cohort 3-5 Hours | Dose Timing Cohort 1-3 Hours
Started | 3 | 3 | 3 | 3 | 3 | 6 | 6
Completed | 3 | 3 | 3 | 3 | 2 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — COVID-19 related hospitalization | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients were accrued into the Dose Defining Cohorts (Dose Escalation/De-Escalation) and the Dose Timing Cohorts using the inclusion and exclusion criteria as defined in the protocol.
Groups:
- Dose Defining 100mg: This arm of the study will include Dose Defining cohort at 100mg. ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 200mg: This arm of the study will include Dose Defining cohort at 200mg. ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 400mg: This arm of the study will include Dose Defining cohort at 400mg. ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 500mg: This arm of the study will include Dose Defining cohort at 500mg. ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 600mg: This arm of the study will include Dose Defining cohort at 600mg. ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing 1-3hrs: This arm of the study will include Dose Timing cohorts of ALM-488 administration 1-3 hrs before surgery.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing 3-5 Hrs: This arm of the study will include Dose Timing cohorts of ALM-488 administration 3-5 hrs before surgery.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Total: Total of all reporting groups
Arm/Group | Dose Defining 100mg | Dose Defining 200mg | Dose Defining 400mg | Dose Defining 500mg | Dose Defining 600mg | Dose Timing 1-3hrs | Dose Timing 3-5 Hrs | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 2 | 3 | 5 | 2 | 20
  >=65 years | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 41 [27 to 56] | 49.7 [31 to 64] | 56.7 [33 to 81] | 68 [60 to 79] | 56.7 [54 to 59] | 36 [20 to 68] | 65 [48 to 75] | 52.6 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 2 | 5 | 2 | 13
  Male | 1 | 2 | 3 | 2 | 1 | 1 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 0 | 0 | 3 | 4 | 5 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2 | 3 | 0 | 0 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Safety - The Number of Patients With ALM-488 Related Adverse Events
Description: The number of patients with ALM-488 related Adverse Events according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: 28 (+5) days
Measure: Count of Participants; unit: Participants
Groups:
- Dose Defining 100mg: This arm of the study will include ALM-488 dose 100mg
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 200mg: This arm of the study will include ALM-488 dose 200mg
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 400mg: This arm of the study will include ALM-488 dose 400mg
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 500mg: This arm of the study will include ALM-488 dose 500mg
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 600mg: This arm of the study will include ALM-488 dose 600mg
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing 1-3hrs: This arm of the study will include ALM-488 timing of administration 1-3 hours before surgery.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing 3-5 Hrs.: This arm of the study will include ALM-488 timing of administration 3-5 hours before surgery.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
Arm/Group | Dose Defining 100mg | Dose Defining 200mg | Dose Defining 400mg | Dose Defining 500mg | Dose Defining 600mg | Dose Timing 1-3hrs | Dose Timing 3-5 Hrs.
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Time of Peak ALM-488 Concentration in Plasma (Cmax)
Description: Time of peak ALM-488 concentration in plasma following intravenous ALM-488 infusion (hours).
Time Frame: 28 (+5) days
Population: Patients were accrued into the Dose Defining Cohorts (Dose Escalation/De-Escalation) and the Dose Timing Cohorts using inclusion and exclusion criteria as specified in the protocol.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Dose Defining 100mg: This arm of the study will include Dose Defining 100mg cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 200mg: This arm of the study will include Dose Defining 200mg cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 400mg: This arm of the study will include Dose Defining 400mg cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 500mg: This arm of the study will include Dose Defining 500mg cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Defining 600mg: This arm of the study will include Dose Defining 600mg cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing 1-3hrs: This arm of the study will include Dose timing of ALM-488 administration 1-3hrs before surgery cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
- Dose Timing 3-5 Hours.: This arm of the study will include Dose timing of ALM-488 administration 3-5hrs before surgery cohort.
  ALM-488: ALM-488 Sterile Solution is an intravenously administered, synthetic, peptide dye conjugate indicated for the real-time intraoperative fluorescence detection and localization of nerve tissue.
Arm/Group | Dose Defining 100mg | Dose Defining 200mg | Dose Defining 400mg | Dose Defining 500mg | Dose Defining 600mg | Dose Timing 1-3hrs | Dose Timing 3-5 Hours.
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6
hours | 0.50 (0.00) | 0.50 (0.00) | 0.50 (0.00) | 0.42 (0.14) | 0.42 (0.14) | 0.42 (0.13) | 0.40 (0.14)

ADVERSE EVENTS:
Time Frame: 28 (+5) days
Groups:
- Dose Defining 100mg: This group of the study will receive 100mg of ALM-488.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.
- Dose Defining 200mg: This group of the study will receive 200mg of ALM-488.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.
- Dose Defining 400mg: This group of the study will receive 400mg of ALM-488.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.
- Dose Defining 500mg: This group of the study will receive 500mg of ALM-488.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.
- Dose Defining 600mg: This group of the study will receive 600mg of ALM-488.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.
- Dose Timing 1-3hrs: This group of the study will receive ALM-488 1-3 hours before surgery.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.usly administered.
- Dose Timing 3-5hrs: This group of the study will receive ALM-488 3-5 hours before surgery.
  Bevonescein (ALM-488): ALM-488 Sterile Solution is an intravenously administered peptide-dye conjugate for nerve visualization during surgery.usly administered.
Arm/Group | Dose Defining 100mg | Dose Defining 200mg | Dose Defining 400mg | Dose Defining 500mg | Dose Defining 600mg | Dose Timing 1-3hrs | Dose Timing 3-5hrs
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 0/3 | 2/3 | 3/6 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Defining 100mg (N=3) | Dose Defining 200mg (N=3) | Dose Defining 400mg (N=3) | Dose Defining 500mg (N=3) | Dose Defining 600mg (N=3) | Dose Timing 1-3hrs (N=6) | Dose Timing 3-5hrs (N=6)
neck infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Defining 100mg (N=3) | Dose Defining 200mg (N=3) | Dose Defining 400mg (N=3) | Dose Defining 500mg (N=3) | Dose Defining 600mg (N=3) | Dose Timing 1-3hrs (N=6) | Dose Timing 3-5hrs (N=6)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
salivary gland fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
non cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
confusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abcess, neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
sialocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04420689/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04420689/SAP_002.pdf